CLINICAL TRIAL: NCT05323136
Title: A Phase 1, Open-Label, Sequential, Adaptive, Single Dose Study to Evaluate the Effects of Renal Impairment on the Pharmacokinetics and Pharmacodynamics of MT1002 for Injection
Brief Title: Evaluate the Effects of Renal Impairment on the Pharmacokinetics and Pharmacodynamics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT1002-I-C02
Record Dates: First submitted 2022-03-26; First posted 2022-04-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: ACS - Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Sequence 1: planned to dose first 1 or 2 sentinels (1 or 2 moderate RI patients) before dosing remaining non-sentinel moderate RI patients. There will be 6 patients with moderate RI in Group 1: RF within 30-59 mL/min. Another group of 6 non-sentinel HVs (Group 2: normal RF, ≥ 90 mL/min) will be one-to-one matched to 6 patients of moderate RI by age, BMI, and gender and may be dosed in parallel to 6 moderate RI patients with same single dose of MT1002.
  Sequence 2: same precaution in Sequence 1 will be used: use of staggered dosing schedule where 1 or 2 sentinel subjects (1 or 2 severe RI patients) will be dosed first before dosing remaining non-sentinel RI patients. There will be 6 patients with severe RI, Group 3: RF < 30 mL/min. A group of up to 6 non-sentinel HVs (normal RF, ≥ 90 mL/min) will be one-to-one matched to 6 patients of severe RI by age, BMI, and gender and will be dosed with same single dose of MT1002.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Renal impairment (Experimental): moderate and severe Renal impairment subjects
  Interventions: Drug: MT1002 for Injection
- Healthy control (Experimental): Healthy control subjects with normal renal function
  Interventions: Drug: MT1002 for Injection

INTERVENTIONS:
Drug: MT1002 for Injection — single dose: 0.90 mg/kg initial loading dose (bolus intravenous injection) over 5 minutes + 1.8 mg/kg/hour (infusion) for 4 hours.

SUMMARY:
The study is a multicenter, Phase 1, open-label, sequential, adaptive, single dose, PK/PD study in subjects with moderate and severe RI and healthy volunteers (HV).

DETAILED DESCRIPTION:
Because MT1002 for Injection is being developed for use as an anticoagulant and antiplatelet in patients with ACS and in patients undergoing PCI, these patients may have impaired RF, and it is important to evaluate whether exposure-response or exposure-safety relationship will be altered in RI. In addition, according to the FDA recommendations, a dedicated RI study including severe RI must be conducted.

The study will be performed in 2 sequences, with interim safety, tolerability, PK, and PD review between both sequences:

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker, ≥ 18 and ≤ 80 years of age, with BMI > 18.0 and < 40.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Female subjects (except for post-menopausal women) must agree to use an adequate method of contraception during the study and for 90 days following the end-of-study visit.
3. Female subjects of non-childbearing potential must be:

   1. Post-menopausal or
   2. Surgically sterile.
4. Male subjects who are not vasectomized for at least 3 months prior to dosing, and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from dosing dose and for 90 days after dosing.
5. Able to understand the study procedures and provide signed informed consent to participate in the study.

   Inclusion Criteria for Subjects with Normal RF (Control Group):
6. Have a RF ≥ 90 mL/min (using the MDRD4 Equation).
7. Healthy as defined by:

   1. The absence of clinically significant illness and surgery within 4 weeks prior to study drug administration.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, cerebrovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
8. Matched to subjects with RI (moderate or severe) according to gender, age (± 10 years), and BMI (± 15%) to the extent possible.

   Inclusion Criteria for Patients with RI:
9. Have a diagnosis of RI that has been stable, without significant change in overall disease status in the last 3 months prior to screening as determined by the PI.
10. Have a RF expressed in mL/min (using MDRD4 Equation) within the range of at screening:

    1. 30 to 59 mL/min (Moderate RI, Group 1);
    2. < 30 mL/min (Severe RI, Group 3) not requiring dialysis.

Exclusion Criteria:

1. Positive pregnancy test at screening or Baseline (Day -1), lactating female subject, or planned to become pregnant during the study.
2. Positive urine cotinine test, alcohol breath test, or drug test, unless for RI patients only, the subject uses any of these drugs as prescriptions that is approved by the PI.
3. Positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody at screening, or active infections.
4. History of significant allergic reactions (e.g., anaphylactic reaction, hypersensitivity, angioedema) to any drug, to mannitol, or to any excipient in the formulation of MT1002 for Injection.
5. Any acute illness within 14 days prior to the screening visit.
6. Clinically significant history of congenital or acquired bleeding disorders, thrombocytopenia or functional platelet defects, gastrointestinal disease with or without active ulceration, active cancer, vascular retinopathy, bronchiectasis, pulmonary cavitation, or pulmonary bleeding.
7. History of major bleeding, trauma, surgical procedure of any type, or vaginal delivery within 6 months prior to screening.
8. Personal or family history of clotting or coagulation disorder or abnormality, thrombovascular disease or any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, anticoagulants or platelet inhibitors.
9. History of peptic ulcer, gastrointestinal bleeding (including hematemesis, melena, rectal bleeding) or bleeding from hemorrhoids within 6 months prior to screening.
10. History of easy bruising, excessive bleeding from an injury or after surgery or dental work, minor bleeding episodes such as epistaxis, rectal or hemorrhoidal bleeding (spots of blood on toilet paper), blood in urine or stool or history of black stools, or gingival bleeding within 3 months prior to screening.
11. Females with a history of dysfunctional uterine bleeding, including history of menorrhagia (heavy or long menstrual bleeding), metrorrhagia or polymenorrhea.
12. PT or aPTT > upper limit of normal at Screening or Day -1.
13. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening or menses) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the dosing.

    Exclusion Criteria for Subjects with Normal RF (Control Group):
14. Clinically significant abnormal laboratory test results (e.g. alanine aminotransferase (ALT), alkaline phosphatase (AP), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT) or bilirubin) as judged by the Investigator or designee at Screening.
15. Clinically significant electrolyte abnormalities (e.g., hypokalemia or hypomagnesemia), congestive heart failure, or other currently prescribed medicinal products that lead to QT prolongation.
16. Administration of any blood product or anticoagulant within 1 month prior to screening.
17. Clinically significant ECG abnormalities (that could have jeopardized the subject's safety to participate in this study or a screening 12-lead ECG that demonstrated any one of the following: HR > 100 beats per minute (bpm), QRS > 120 msec, QTcF ≥450 ms in males or ≥470 ms in females, or PR > 220 msec, or vital signs abnormalities (systolic BP lower than 90 or over 140 mmHg, diastolic BP lower than 50 or over 90 mmHg, HR less than 50 or over 100 bpm, or RR less than 10 or over 22 bpm) at screening.

    Exclusion Criteria for Patients with Impaired RI (Moderate and Severe Impairment):
18. Unstable medical conditions or acute exacerbation of renal disease within 14 days of study drug administration.
19. Fluctuating or rapidly deteriorating RF as indicated by recent history or worsening of clinical and/or laboratory signs of RI as judged by the PI.
20. History, symptoms, or signs of severe hepatic impairment.
21. Subject who has renal disease secondary to malignancy.
22. Subjects with acute renal failure.
23. Subjects requiring dialysis.
24. Evidence of significantly impaired organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiogram (ECG) or clinical laboratory determinations beyond what is consistent with the target population.
25. Subject is excluded at the discretion of the PI with consultation with the Medical Monitor if any of the following laboratory parameters at Screening and/or Baseline (Day -1) are above the followings: total bilirubin (TBL) > 1.5 × ULN, ALT and AST > 2 × ULN and ALP > 3 × ULN) at Screening or Day -1; hemoglobin < 8.5 g/dL.
26. Clinically significant ECG abnormalities or vital sign abnormalities (systolic BP lower than 90 or over 160 mmHg, diastolic BP lower than 50 or over 110 mmHg, or HR less than 45 or over 100 bpm) at screening. Any BP and HR values can be repeated at the discretion of the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Plasma PK | 24 hour
  plasma AUC0-t value
Plasma PK | 24 hour
  plasma AUC0-inf value
plasma PK | 24 hour
  plasma Cmax value
plasma PK | 24 hour
  plasma Tmax
plasma PK | 24 hour
  plasma T½ el value
Urine PK | 24 hour
  urine Ae0-t value
Urine PK | 24 hour
  Urine Rmax value
Urine PK | 24 hour
  Urine TRmax value
Urine PK | 24 hour
  Urine Clr value

SECONDARY OUTCOMES:
Adverse events | 30 days
  AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Panax Clinical Research, LLC., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No